CLINICAL TRIAL: NCT03180450
Title: The Study of Heart Failure With Human Umbilical Cord Mesenchymal Stem Cells (hUC-MSC)
Brief Title: The Study of Heart Failure With Human Umbilical Cord Mesenchymal Stem Cells (19#iSCLife®-HF)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-IMIMH-04
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Human Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): conventional treatment; Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#) by i.v.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#); Drug: conventional treatment
- Control group (Placebo Comparator): Conventional treatment
  Interventions: Drug: conventional treatment

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#) — Allogeneic umbilical cord mesenchymal stem cells will transfusion by intravenous transplantation.
  Arms: Treatment group
Drug: conventional treatment — The drug and usage will be determined based on patient's condition, including milrinone, furosemide, beta-blocker blues, Angiotensin-Converting Enzyme Inhibitors (ACEI), angiotension receptor blocker (ARB), or antiplatelet aggregation etc.

SUMMARY:
The purposes of the study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cells (hUC-MSC) in treating heart failure patients

DETAILED DESCRIPTION:
This is a randomized, paralleled study. Patients will be divided into two groups of treatment and control. all of them will receive conventional treatment based on specific condition, including digitalis, milrinone, furosemide, beta-blocker blues, Angiotensin-Converting Enzyme Inhibitors (ACEI), angiotension receptor blocker (ARB), and antiplatelet aggregation etc. Treatment group patients will receive hUC-MSC. Follow-up visit will occur on 3 months, 6 months, and 12 months after the cell transfusion. Vital signs, blood routine test, urine routine test, liver function examination, etc, will be placed to evaluate the safety of hUC-MSC treatment. And the change of symptoms to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate in clinical trial, and sign informed consent form
* with cardiac failure symptoms, including oppression in chest, breathe hard, lower limb edema. And new york heart association class as two to four
* heart color ultrasound indicate left ventricular ejection fraction (LVEF) < 40%
* content of serum NT-proBNP > 450pg/ml

Exclusion Criteria:

* with severe drug allergy history or allergic constitution
* patients were severe infected
* with malignant tumor or with high tumor marker
* with severe cardiorespiratory dysfunction, hematological system disease
* with severe mental disorder, cognitive impairment
* with persistent atrial fibrillation, valvular heart disease, dilated cardiomyopathy, hypertrophic cardiomyopathy or restrictive cardiomyopathy patients
* end-stage renal insufficiency, pregnancy, or breast feeding women
* bleeding tendency, active gastrointestinal ulcer
* recent have major surgery, stroke, cancer, hepatic function insufficiency or other life-threatening condition.
* under other therapy that possibly influence MSC security or efficacy
* donor: HIV, active hepatitis B/C infection, Syphilitic antibody positive
* participant/donor: alcoholism, drug addicted, mental disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart color ultrasound evaluation | 12 months
  Criteria:
  * Excellent: ejection fraction improve to > 50%;
  * Efficient: ejection fraction improved;
  * Inefficient: ejection fraction same as before treatment;
  * Exacerbation: ejection fraction declined.

SECONDARY OUTCOMES:
Single therapy effectiveness evaluation | 12 months
  Evaluate criteria:
  * Recovery: symptoms disappear
  * Excellent: symptoms improved obviously
  * Efficient: symptoms improved
  * Inefficient: symptoms no change or worse

CONTACTS AND LOCATIONS:
Overall Officials: Nashundalai, Study Director — Inner Mongolia International Mongolian Hospital; Lei Guo, Dr., Study Chair — China-Japan Union Hospital, Jilin University
Locations (1):
- Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No